CLINICAL TRIAL: NCT03745924
Title: A Non-Interventional Post-Authorisation Safety Study (PASS) in Male Haemophilia B Patients Receiving Nonacog Beta Pegol (N9-GP) Prophylaxis Treatment
Brief Title: A Study Following Males With Haemophilia B on Prophylaxis With Refixia/REBINYN
Status: Enrolling by invitation | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN7999-4031; U1111-1165-8657 (Other: World Health Organization (WHO)); EUPAS26592 (Registry Identifier: EU PAS Register)
Record Dates: First submitted 2018-11-15; First posted 2018-11-19 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Haemophilia B
MeSH Terms: conditions — Hemophilia B | interventions — nonacog beta pegol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with haemophilia B: Patients with haemophilia B without current inhibitors
  Interventions: Drug: Nonacog beta pegol

INTERVENTIONS:
Drug: Nonacog beta pegol — Participants are treated with commercially available nonacog beta pegol (N9-GP) according to local clinical practice at the discretion of the treating physician

SUMMARY:
This study will collect information on side effects and how well Refixia/REBINYN works during long-term treatment (prophylaxis) in males with haemophilia B. While taking part in this study, participants will receive the same treatment as given to them by their study doctor. All visits at the clinic are done in the same way as the participants are used to. During visits at the clinic, participants might be asked for some relevant tests if considered useful by their study doctor. During the visits, the participants study doctor might ask if the participants had any side effects since their last study visit. The participants will be asked to note down the number of bleeds and the treatment of their bleeds as well as their regular prophylaxis. During the visits to the clinic, the participants will be asked to answer some questionnaires about their quality of life and their ability to be physically active. The participant's participation in the study will last for 4-9 years, depending on when they join the study. Participants are free to leave the study at any time and for any reason. This will not affect their current and future medical care.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent obtained before any study-related activities (study-related activities are any procedure related to recording of data according to the protocol).
* Male patients at any age with haemophilia B assigned to N9-GP prophylaxis treatment
* Decision to initiate treatment with commercially available N9-GP has been made by the patient(s)/Legally Authorised Representative(s) (LAR(s)) and the treating physician before and independently from the decision to include the patient in this study

Exclusion Criteria:

* Previous participation in this study. Participation is defined as signed informed consent
* Known or suspected hypersensitivity to N9-GP or related products
* Mental incapacity, unwillingness or language barriers precluding adequate understanding or cooperation
* Clinical suspicion or presence of FIX inhibitor at time of inclusion.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with haemophilia B
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2027-12-15 (Estimated); Study Completion 2027-12-15 (Estimated)

PRIMARY OUTCOMES:
Number of Adverse Drug Reactions (ADRs) (FIX inhibitors, allergic reactions, and thromboembolic events) | From start of study period (week 0) to end of study period (up to 9 years)
  Count of events

SECONDARY OUTCOMES:
Number of Serious Adverse Events (SAEs) | From start of study period (week 0) to up to 9 years
  Count of events
Number of bleeding episodes during long-term routine use of N9-GP (prophylaxis) as assessed by annualised bleeding rate (ABR) | From start of study period (week 0) to up to 9 years
  Count of episodes
Number of treatment requiring bleeding episodes during long-term routine use of N9-GP (prophylaxis) as assessed by annualised bleeding rate (ABR) | From start of study period (week 0) to up to 9 years
  Number of episodes
Haemostatic effect of N9-GP when used for treatment of bleeding episodes | From start of study period (week 0) to up to 9 years
  Count of bleeding episodes. Haemostatic effect is assessed as success/failure based on a four-point scale for haemostatic response (excellent, good, moderate and poor) by counting excellent and good as success and moderate and poor as failure
Haemostatic response of N9-GP when used in perioperative management | From start of study period (week 0) to end of study period (up to 9 years)
  Count of bleeding episodes. Haemostatic response is assessed as success/failure based on a four-point scale for haemostatic response (excellent, good, moderate and poor) by counting excellent and good as success and moderate and poor as failure

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Reporting Anchor and Disclosure (1452), Study Director — Novo Nordisk A/S
Locations (28):
- AKH - Klin. Abt. f. Haematologie u. Haemostaseologie, Vienna, Austria
- Belgium (3):
  - Cliniques universitaires Saint-Luc - Service Hématologie, Brussels
  - UZ Antwerpen - UZA - Kinderhemato-Oncologie, Edegem
  - UZ Leuven - Hart en Vaatziekten, Leuven
- Canada (7):
  - University of Calgary Cumming School of Medicine, Calgary, Alberta
  - Univ of Alberta Hospital Res, Edmonton, Alberta
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Health Science Centre, St. John's, Newfoundland and Labrador
  - Hamilton Health Sciences Corp, Ontario, Hamilton, Ontario
  - Hamltn Hth Sci/McMstr Child Hosp, Hamilton, Ontario
  - The Hospital for Sick Children, Toronto, Ontario
- KBC Zagreb, Rebro, Hemofilija centar, Zagreb, Croatia
- Czechia (2):
  - FN Brno odd. hematologie, Brno
  - Fakultni nemocnice Plzen - Lochotin, Pilsen
- Skejby Blodsygdomme, blødercentret, Aarhus N, Denmark
- Helsinki University Central Hospital/Coagulation Disorder Un, Helsinki, Finland
- Germany (2):
  - Vivantes Netzwerk für Gesundheit GmbH - Vivantes Klinikum im Friedrichshain, Berlin
  - Universitätsklinikum Bonn - Institut für Experimentelle Hämatologie, Bonn
- Greece (2):
  - "Laiko" General Hospital of Athens, Athens
  - Aghia Sophia Childrens' Hospital, Athens
- Klinisk forskningspost, Oslo, Norway
- Portugal (2):
  - Hospital São José, Lisbon
  - Unidade Local de Saúde São José EPE- Hospital D. Estefânia, Lisbon
- Universitätsspital Zürich - Klinik für Medizinische Onkologie und Hämatologie, Zurich, Switzerland
- United Kingdom (4):
  - Aberdeen Royal Infirmary - Haematology, Aberdeen
  - University Hospital of Wales - Haemophilia, Cardiff
  - Royal Manchester Children's Hospital, Manchester
  - Royal Hallamshire Hospital, Sheffield

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com